CLINICAL TRIAL: NCT03134846
Title: Image Guided Surgery for Margin Assessment of Head and Neck Cancer Using Cetuximab-IRDye800CW cONjugate
Acronym: ICON
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Collaborators: UMC Utrecht (Other); Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, dr. M.J.H. Witjes, MD, PhD, University Medical Center Groningen
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: NL58585.042.16
Record Dates: First submitted 2017-04-20; First posted 2017-05-01 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Margin Assessment
Keywords: Intraoperative fluorescence imaging; Cetuximab-IRDye800CW; Molecular imaging
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Intervention Model Description: Phase 1: 3x3 Dose-escalation with 3 different doses Cetuximab-IRDye800CW Phase 2: Prospective cross sectional diagnostic study. After having established the optimal cetuximab-IRDye800CW dose we will extent the study by including up to 70 patients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Phase 1: 10mg Cetuximab-IRDye800CW (Experimental): Three patients will receive 10mg Cetuximab-IRDye800cv I.V. four days prior to surgery.
  Interventions: Drug: Cetuximab-IRDye800CW
- Phase 1: 25mg Cetuximab-IRDye800CW (Experimental): Patients will receive 25mg Cetuximab-IRDye800cv I.V. four days prior to surgery.
  Interventions: Drug: Cetuximab-IRDye800CW
- Phase 1: 50 mg Cetuximab-IRDye800CW (Experimental): Patients will receive 50mg Cetuximab-IRDye800cv I.V. four days prior to surgery.
  Interventions: Drug: Cetuximab-IRDye800CW
- Phase 1: 75mg cetuximab + 15 mg Cetuximab-IRDye800CW (Experimental): Patients will receive 75mg cetuximab + 15 mg Cetuximab-IRDye800CW I.V. four days prior to surgery.
  Interventions: Drug: Cetuximab-IRDye800CW
- Phase 1: 75mg cetuximab + 25 mg Cetuximab-IRDye800CW (Experimental): Patients will receive 75mg cetuximab + 25 mg Cetuximab-IRDye800CW I.V. four days prior to surgery.
  Interventions: Drug: Cetuximab-IRDye800CW
- After having established the optimal cetuximab-IRDye800CW dose (Experimental): After having established the optimal cetuximab-IRDye800CW dose we will extent the study by including up to 70 patients for this specific dose (as determined in phase 1).
  Interventions: Drug: Cetuximab-IRDye800CW

INTERVENTIONS:
Drug: Cetuximab-IRDye800CW — Pre-operatively administration of Cetuximab-IRDye800CW for intra operative margin assessment using a fluorescent antibody-based optical tracer
  Other Names: Cetuximab-800cw

SUMMARY:
Surgery remains a main pillar in the treatment of head and neck squamous cell carcinoma (HNSCC). The margin status is the main prognostic factor of local tumor control in surgically treated HNSCC and will determine the postoperative treatment strategy. A margin of ≤1 mm of normal tissue is considered a positive margin and requires either a re-operation or postoperative chemoradiation with a combination of cisplatin and 5-FU, which substantially increases morbidity. Margins wider than 1 mm but less than 5 mm require re-operation, or, if that is not possible, post-operative radiotherapy without the concomitant use of chemotherapy. Currently, no technology is available in the operating room, which reliably supports tumor excision in terms of margin status. In fact, surgeons can only combine pre- operative imaging data with tactile and visual information during surgery for assessing tumor margins with limited accuracy. With the introduction of molecular imaging techniques using near infrared (NIR) fluorescent optical contrast agents coupled to targeted compounds, new avenues have opened up for intra-operative assessment of tumor margins. Tracers are based on antibodies directed against Vascular Endothelial Growth Factor-A, i.e. bevacizumab-IRDye800CW, in patients with breast cancer or against Epidermal Growth Factor Receptor, i.e. cetuximab-IRDye800CW, in patients with HNSCC. First trials have shown that systemic administration of these compounds is safe and tumor specific. These findings prompted us to design this innovative application in a clinical trial for the intraoperative assessment of tumor margins during surgical treatment of HNSCC using cetuximab-IRDye800CW.

DETAILED DESCRIPTION:
Surgery remains a main pillar in the treatment of head and neck squamous cell carcinoma (HNSCC). The margin status is the main prognostic factor of local tumor control in surgically treated HNSCC and will determine the postoperative treatment strategy. A margin of ≤1 mm of normal tissue is considered a positive margin and requires either a re-operation or postoperative chemoradiation with a combination of cisplatin and 5-FU, which substantially increases morbidity. Margins wider than 1 mm but less than 5 mm require re-operation, or, if that is not possible, post-operative radiotherapy without the concomitant use of chemotherapy. Currently, no technology is available in the operating room, which reliably supports tumor excision in terms of margin status. In fact, surgeons can only combine pre- operative imaging data with tactile and visual information during surgery for assessing tumor margins with limited accuracy. With the introduction of molecular imaging techniques using near infrared (NIR) fluorescent optical contrast agents coupled to targeted compounds, new avenues have opened up for intra-operative assessment of tumor margins. Tracers are based on antibodies directed against Vascular Endothelial Growth Factor-A, i.e. bevacizumab-IRDye800CW, in patients with breast cancer or against Epidermal Growth Factor Receptor, i.e. cetuximab-IRDye800CW, in patients with HNSCC. First trials have shown that systemic administration of these compounds is safe and tumor specific. These findings prompted us to design this innovative application in a clinical trial for the intraoperative assessment of tumor margins during surgical treatment of HNSCC using cetuximab-IRDye800CW. The study is subsidized by the Dutch Cancer Foundation.

Objectives The main purpose is to establish the intraoperative use of cetuximab-IRDye800CW as a reliable marker for residual tumor in resection margins after surgical removal of HNSCC. The objective is to establish the positive predictive value of cetuximab-IRDye800CW fluorescence as a marker for a tumor positive resection margin.

Study design The study is designed as a phase 1-2, single center prospective cross sectional diagnostic study in patients with HNSCC that require surgical excision. First, a dose finding study will be performed in 9 patients using 10, 25 and 50 mg of cetuximab-IRDye800CW with three patients per dose cohort. In the first and only performed study at the University of Alabama (UAB) using cetuximab-IRDye800CW in the visualization of HNSCC, the dose found to be optimal was 25mg/m2. We therefore think that a sufficient dose will be found within the proposed range. The most optimal dose from the three studied doses will be used in the second part of the study which will include a cohort of 70 patients. The choice of cetuximab-IRDye800CW dose will be a balance between the lowest dose vs. a clinically usable tumor to background ration (TBR) on the fluorescence images.

During the second phase of the study tumor margins will be studied in a cohort of 70 patients to determine the positive predictive value of optical imaging to identify positive margins. Based on historical data retrieved from our HNSCC database at UMCG we anticipate in a cohort of 70 patients at least 14 (20%) margin-positive patients and a 90% EGFR overexpression rate. We anticipate a sensitivity of 90% of the cetuximab-IRDye800CW conjugate based on the EGFR overexpression rate, which we will be able to measure with sufficient precision ( 95%CI of 60-96%).

Study population Patients eligible for inclusion should suffer from a squamous cell carcinoma in the head and neck region (HNSCC) of which the head and neck tumor board of the UMCG has advised to be treated by surgical removal.

Patient related study procedures Tracer administration: patients will visit the hospital four days prior to the planned surgery of their HNSCC. The cetuximab-IRDye800CW will be injected by slow infusion and patients will be monitored for potential side effects. The dose will be either 10, 25 or 50 mg of cetuximab-IRDye800CW which is less or equal to 10% of the dose of cetuximab when used for curative treatment of HNSCC (usually 400mg/m2 loading dose and 250mg/m2 maintenance dose).

Pre-operative fluorescence imaging, spectroscopy and assessment of tracer concentration/stability Only during phase 1, patient will undergo pre-operative imaging and spectroscopy measurement one day prior to surgery. Furthermore, 6 blood samples will be drawn and tissue will be collected at different time point during the study for assessment of tracer concentration/stability.

Intraoperative fluorescence imaging and spectroscopy Study aims: The aim is to identify squamous cell carcinoma as fluorescent spots in the margin of a tumor resection specimen or in the wound bed in the patient.

Parameters: Fluorescence imaging and spectroscopy: Fluorescence images will provide an overview of where cetuximab-IRDye800CW fluorescence is located in the resection specimen and the wound bed in the patients. The intra operative camera is very sensitive for cetuximab-IRDye800CW fluorescence. One drawback is that on the fluorescence image the exact depth from which the fluorescence signal is generated cannot be established. Furthermore, most likely there will be background fluorescence signals from normal tissue. Therefore, confirmation of the fluorescence signal on images requires quantification of the fluorescence signal. This can be performed by using a spectroscopy technique (MDSFR spectroscopy) that can quantify (in M/m3) specifically IRDye800CW-fluorescence by placing a fiber tip in contact with the tissue. This spectroscopy technique has a shallow sampling depth of 1-2 mm. If fluorescence is generated from deeper layers, the signal of spectroscopy will be low (only background signal from muscle, connective tissue and salivary glands). If the IRDye800CW-fluorescence signal is generated from tumor in the resection margin the fluorescence signal will be much higher because SCC-tumor cells overexpress EGFR. The parameter that will be established is the threshold level at which background cetuximab-IRDye800CW spectroscopy signal can be separated from much higher spectroscopy signals of cetuximab-IRDye800CW accumulated in tumor.

Pathology: The tumor specimen will be processed for histology according to the current standard used in clinical cancer care. Diagnosis on margins, selected histological features necessary for clinical decision making will be provided. Next to this fluorescence images will be collected from the tumor specimen and biopsies. Margin width and number of positive margins will be noted and correlated to the location of fluorescent locations in the margins. From this positive predictive value will be calculated.

Burden, risks and benefit related to participation Burden - Time investment: Patients need to make one extra visit to the UMCG four days before their planned surgery that will take approximately 2 hours. Usually patients are admitted one day prior to the planned surgery. Therefore the measurements one day before surgery will not require extra time investment Burden-extra procedures: 1) Intravenous administration of cetuximab-IRDye800CW. 2) Fluorescence images will be taken from the tumor one day prior to surgery in the first cohort of nine patients. 3) The estimated time for taking fluorescence images and spectroscopy measurements is approximately 30min. Therefore the time under general anesthesia will be prolonged. The usual time of surgical procedures for removal of HNSCC ranges from 2 hours to 15 hours, depending on complexity of the surgical procedure. 4) from the wound bed in the patient that exists after tumor excision, biopsies will be taken in the ongoing general anesthesia, of spots positive of cetuximab-IRDye800CW as seen on the fluorescence imaging and confirmed by spectroscopy.

Risks: Allergic reactions to cetuximab have been reported but this is considered a low risk. No preclinical or clinical study reported higher than grade 2 adverse events. the first study with cetuximab-IRDye800CW no serious events were reported in six patients.

Benefit: Patients will have no benefit from this study directly. Surgery will be planned as usual. During surgery, no decisions will be made based on the fluorescence imaging. The benefit of this study will be the establishment of usefulness of cetuximab-IRDye800CW during surgery to identify margins containing tumors. The results of these types of study will be at least beneficial for other patients with cancer in the future. Clinical experience will be obtained with fluorescent labeled antibody in intra operative margin assessment during surgery of HNSCC.

ELIGIBILITY:
Inclusion criteria

1. Biopsy confirmed diagnosis of primary or recurrent HNSCC and scheduled to undergo surgical resection as decided by the Multi-Disciplinary Head and Neck Tumor Board of the UMCG.
2. Age ≥ 18 years
3. Written informed consent
4. Adequate potential for follow up
5. Acceptable hematologic status, kidney function, and liver function, as standard surgery protocol requires.

Exclusion criteria

1. Medical or psychiatric conditions that compromise the patient's ability to give informed consent
2. Concurrent uncontrolled medical conditions.
3. Received an investigational drug within 30 days prior to the dose of cetuximab-IRDye800CW
4. Tumors at sites of which the surgeon would assess that in vivo imaging would not be feasible
5. Had within 6 months prior to enrollment: myocardial infarction, cerebrovascular accident, uncontrolled cardiac heart failure, significant liver disease, unstable angina
6. Inadequately controlled hypertension with or without current antihypertensive medications.
7. History of infusion reactions to cetuximab or other monoclonal antibody therapies
8. Pregnant or lactating women. Documentation of a negative pregnancy test must be available for women of childbearing potential. Woman of childbearing potential are premenopausal women with intact reproductive organs and women less than two years after menopause.
9. Evidence of QT prolongation on pretreatment ECG (greater than 440 ms in males or greater than 450 ms in females)
10. Lab values that in the opinion of the primary surgeon would prevent surgical resection.
11. Patients receiving Class IA (quinidine, procainamide) or Class III (dofetilide, amiodarone, sotalol) antiarrhythmic agents.
12. Magnesium, potassium and calcium lower than the lower limit of normal range.
13. Life expectancy < 12 weeks
14. Karnofsky performance status < 70%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Estimated)
Dates: Start 2017-12-16 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Determine the optimal dose of Cetuximab-IRDye800CW for imaging | Five months
  The primary endpoint for the feasibility study (9 patients) will be confirmation of the clinically applicable dose of cetuximab-IRDye800CW. The aim is to obtain at least a TBR higher than 2 by fluorescence imaging with the intra operative camera. This number has been found to give sufficient demarcation of tumor to normal tissue on wide field images.
Phase 2: Threshold level of fluorescence | Three years
  Determine a threshold level of fluorescence that can discriminate between EGFR distribution in normal tissue and a margin with EGFR-positive tumor.

SECONDARY OUTCOMES:
Phase 1: Secondary outcome: Safety | Five months
  Adverse events will be monitored
Phase 1: Secondary outcome: Identification of positive margins | Five months
  By ex vivo imaging and MDSFR spectroscopy of the excised specimen
Phase 1: Tissue specificity of IRDye800cw | Five months
  Identification of the tissues that show IRDye800CW-fluorescence in the surgical wound bed after tumor removal
Phase 1: Histological location of IRDye800cw | Five months
  Localisation patterns of cetuximab-IRDye800CW in the tumor and normal tissue by microscopy
Phase 2: Secondary outcome: Minimal thickness of the non-fluorescent margin | Three years
  The assessment of the minimal thickness of the non-fluorescent margin of the excised specimen with histopathology and fluorescence microscopy. This will provide us the first data on the relationship between margin thickness when fluorescence cannot be detected.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] de Wit JG, Vonk J, Voskuil FJ, de Visscher SAHJ, Schepman KP, Hooghiemstra WTR, Linssen MD, Elias SG, Halmos GB, Plaat BEC, Doff JJ, Rosenthal EL, Robinson D, van der Vegt B, Nagengast WB, van Dam GM, Witjes MJH. EGFR-targeted fluorescence molecular imaging for intraoperative margin assessment in oral cancer patients: a phase II trial. Nat Commun. 2023 Aug 16;14(1):4952. doi: 10.1038/s41467-023-40324-8. PMID 37587149